CLINICAL TRIAL: NCT01341977
Title: Safety and Efficacy of an Investigational Multi-Purpose Disinfecting Solution (MPDS)
Brief Title: Safety and Efficacy of an Investigational Multi-Purpose Disinfecting Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: C-09-026
Record Dates: First submitted 2009-12-09; First posted 2011-04-26 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2011-09

CONDITIONS: Healthy Contact Lens Wearers
Keywords: Contact Lenses; Contact Lens Care; Multi-Purpose Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcon MPDS (Experimental): Alcon Multi-Purpose Disinfecting Solution (MPDS)
  Interventions: Device: Alcon MPDS
- ReNu Fresh Multi-Purpose Solution (Active Comparator): ReNu Fresh Multi-Purpose Solution
  Interventions: Device: ReNu Fresh MPS

INTERVENTIONS:
Device: Alcon MPDS — Multi-Purpose Solution intended for use with silicone hydrogel and soft contact lenses
  Other Names: Alcon Multi-Purpose Disinfecting Solution (MPDS)
  Arms: Alcon MPDS
Device: ReNu Fresh MPS — ReNu Fresh MPS is a marketed product indicated for cleaning, removing protein deposits, rinsing, disinfecting and storage of soft contact lenses.
  Other Names: ReNu Fresh Multi-Purpose Solution (MPS)
  Arms: ReNu Fresh Multi-Purpose Solution

SUMMARY:
The purpose of this study is to determine if Alcon MPDS is safe and effective for silicone hydrogel and soft hydrogel contact lens wearers.

DETAILED DESCRIPTION:
The purpose of this study is to determine if Alcon Multi-Purpose Disinfecting Solution (MPDS) is safe and effective for silicone hydrogel and soft hydrogel contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Silicone hydrogel or soft contact lens wearers who wear their lenses daily wear (i.e. disinfect lenses every night).
* Patient must be able to read.
* Vision correctable to 20/30 or better with contact lenses.

Exclusion Criteria:

* Sensitivity to multi-purpose solutions.
* Using any topical ocular OTC or prescribed topical ocular medications.
* History or current ocular infections or ocular inflammatory events.
* Ocular surgery within the past year.
* With a medical condition or using medications that cause ocular side effects.
* Participation in any investigational study within the past 30 days.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie M Lemp, MS, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ReNu Fresh Multi-Purpose Solution: ReNu Fresh Multi-Purpose Solution (MPS)
Period: Overall Study
Arm/Group | Alcon MPDS | ReNu Fresh Multi-Purpose Solution
Started | 288 | 285
Completed | 274 | 270
Not Completed | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcon MPDS | ReNu Fresh Multi-Purpose Solution | Total
Number analyzed (Participants) | 288 | 285 | 573
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 23 | 31
  Between 18 and 65 years | 279 | 257 | 536
  >=65 years | 1 | 5 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10.7) | 33.9 (11.4) | 33.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 197 | 411
  Male | 74 | 88 | 162
Region of Enrollment [Number; unit: participants]
  United States | 288 | 285 | 573

OUTCOME MEASURES:

1. Primary Outcome: Subjective Acceptance
Description: Lens Moisture Subject Rated Likert Item (1-Strongly Agree to 5-Strongly Disagree)
Time Frame: Day 90
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcon MPDS | ReNu Fresh Multi-Purpose Solution
Number analyzed (Participants) | 288 | 285
units on a scale | 1.9 (.8) | 2.1 (1.0)

ADVERSE EVENTS:
Time Frame: AE Forms document adverse events during study(occurring after exposure to test article), causality assessment performed by investigator/sponsor. A SAE Form completed & forwarded to Alcon/IRB/EC 24 hours of investigator's knowledge of event
Description: AE Forms document all AEs that occur during study (occurring after exposure to test article), causality assessment performed by investigator/sponsor. A SAE Form completed for all SAEs, forwarded to Alcon/IRB/EC within 24 hours of the investigator's knowledge of the event according to their requirements.
Arm/Group | Alcon MPDS | ReNu Fresh Multi-Purpose Solution
Serious Adverse Events (participants affected / at risk) | 0/288 | 1/285
Other Adverse Events (participants affected / at risk) | 0/288 | 0/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alcon MPDS (N=288) | ReNu Fresh Multi-Purpose Solution (N=285)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — Unrelated to Test Article

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data and discoveries arising out of the Study shall be the sole property of Alcon or its designated affiliate. Alcon reserves the right of prior review of any publication or presentation of the information related to the Study.